CLINICAL TRIAL: NCT06744530
Title: Cardiac RadiothErapy for VEntricular Tachycardia II - a Prospective Observational Cohort Study
Brief Title: Cardiac RadiothErapy for VEntricular Tachycardia II
Acronym: CREVET II
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S69812
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Ventricular Tachycardia (VT)
Keywords: ventricular tachycardia; STAR; Stereotactic radiotherapy
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: stereotactic radiotherapy ablation — Single dose of 25 Gy up to 32.5 Gy on the myocardium in patients with therapy-refractory ventricular tachycardia
  Other Names: STAR; stereotactic body radiotherapy

SUMMARY:
Steoreotactic therapy radioablation has become a standard of care option for patients with therapy-refractory ventricular tachycardia, yet long-term outcome is lacking. The objective of this study is to evaluate the long-term outcomes, both efficacy and safety, after STAR in patients with therapy-refractory ventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for STAR for therapy-refractory VT based on a multidisciplinary discussion
* Ability to give a written informed consent and willingness to return for follow-up

Exclusion Criteria:

* Contra-indications for STAR, including pregnancy or breastfeeding, previous radiotherapy with cardiac involvement, life-expectancy < 6 months in the absence of VT
* Any condition that is deemed a contraindication in the judgment of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with therapy-refractory ventricular tachycardia who are scheduled for stereotactic radiotherapy ablation (STAR) are eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Change in VT burden | 48 months
  Change in VT burden, measured as the frequency of appropriate ICD interventions or documented VT episodes over a 48-month follow-up period. The ICD interrogations are part of standard of care and the majority of patients are included in remote monitoring which automatically sends new VT episodes to the telemonitoring team. The efficacy of STAR will be assessed by analysing both the total VT burden, but also time to first VT event (with and without a 6 week blanking period).

SECONDARY OUTCOMES:
Quality of Life | Baseline and at each follow-up moment: 1 month, 2 months, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months
  The 36-Item Short Form Survey (SF-36) is a set of generic, coherent, and easily administered quality of life measures that rely on patient self-reporting. The SF-36 evaluates 8 domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scale values for each domain range from 0 to 100 where the higher score defines a more favorable health state over a 48-month follow-up period.
All-cause mortality | 48 months
  Survival will be tracked during the 48-month follow-up period. In case of mortality, the cause of death will be registered.
Radiotherapy toxicity | 48 months
  The tolerable acute toxicity rate is defined as a 30-days follow-up without treatment-related grade ≥ 3 adverse events. Late toxicity is defined as toxicity occurring after at least 30 days after the radiation treatment. Toxicity will be assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Left ventricular function | Baseline and at each follow-up moment: 1 month, 2 months, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months
  Left ventricular function on transthoracic echocardiogram (TTE) by measuring left ventricular ejection fraction.
Evolution of valve disease | Baseline and at each follow-up moment: 1 month, 2 months, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months
  Change of pre-existing or new valve stenosis and insufficiency expressed as grade 0 / I / II / III / IV on transthoracic echocardiogram (TTE).
Change of coronary artery disease | Baseline, 2 years and 4 years
  Presence and extent of coronary artery disease on CT coronary angiogram at 2 and 4 years follow-up using the calcium score and CAD-RADs stage.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided